CLINICAL TRIAL: NCT03950037
Title: An Open-label Non-randomized Phase IIa Trial to Evaluate Safety of Early Intervention in Asymptomatic Subarachnoid Neurocysticercosis
Brief Title: SANCC: Clinical Trial Early Intervention
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to complete due to SARS-CoV-2 pandemic
Sponsor: Oregon Health and Science University (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Seth E O'Neal, MD MPH, Assistant professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00019627; 1R01NS103623-01A1 (NIH)
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Subarachnoid Neurocysticercosis
MeSH Terms: interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical intervention (Experimental): Participants are hospitalized for 15-30 days while they receive the antiparasitic drug albendazole along with supportive drugs including dexamethasone and omeprazole.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — Albendazole; 15 mg/k/d divided in two doses (morning and evening), for 30 days, with a ceiling in 1200 mg/d.

SUMMARY:
Subarachnoid neurocysticercosis (SANCC) is a severe infection of the brain by the tapeworm Taenia solium. People who have this infection are usually diagnosed late in the disease process leading to very poor prognosis. This trial studies the safety of early medical intervention in people who have SANCC but do not have symptoms. The trial will enroll 18 participants in Peru.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the risk of serious adverse events (SAE) related to intervention in asymptomatic SANCC; these include drug-related side effects, moderate/severe intracranial hypertension, hydrocephalus requiring shunting or endoscopy, stroke, status epilepticus, or unexplained death.

OUTLINE:

Participants will be hospitalized for approximately 15-30 days while they receive treatment with the antiparasitic drug albendazole, as well as additional drugs (dexmathesaone and omeprazole) to address potential treatment complications. Participants will have continuous monitoring for adverse events while in the hospital. After participants are released to home, they will monitored for adverse events for an additional 12 months through home visits, telephone contact, and monthly clinical evaluations with serologic and radiologic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals older than two years with a diagnosis of asymptomatic SANCC confirmed by MRI.
* SANCC limited to the basal cisterns, the interhemispheric brain space, brain fissures or spine.
* Baseline laboratory results within acceptable ranges (specifically defined in the study protocol)
* Willingness to accomplish the two-week minimum hospitalization required.

Exclusion Criteria:

* Individuals who only have subarachnoid lesions in the convexity of the brain hemispheres will not be included because these lesions commonly respond well to therapy and behave as intraparenchymal lesions
* Co-occurrence of a) more than 20 intraparenchymal lesions in addition to their subarachnoid disease, or b) intraparenchymal lesions greater than 3.0 cm of diameter
* Individuals for whom a surgical intervention to treat their subarachnoid disease is considered clearly superior to a medical intervention
* Previously diagnosis or treatment for cysticercosis.
* Active pulmonary tuberculosis evidenced by chest X-ray and positive sputum smears, or symptoms compatible with tuberculosis (fever+sweats or fever+cough) not otherwise explained
* Individuals with positive markers for active hepatitis
* Other systemic disease that may affect therapy or short-term prognosis, including but not limited to chronic renal failure, hepatic insufficiency, cardiac failure, or steroid-dependent immune diseases
* Pregnancy. If a participant becomes pregnant during the study, she will continue in the study but will have radiological exams delayed until after delivery
* History of hypersensitivity to ABZ
* Chronic alcohol or drug abuse as defined in the study protocol
* Unwilling or unable to provide MRI exams (e.g. patients with ferromagnetic implants)
* Inability or unwillingness of subject or legal representative to give written informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Safety; severe adverse events | The 3 month period directly following the intervention
  Proportion of subjects that experience any severe adverse event that is directly related to the treatment intervention

SECONDARY OUTCOMES:
Safety; all adverse events | The 12 month period directly following the intervention
  Frequency and type of all adverse events
Diagnostic; antigen levels | Months 3,6,9, and 12 after intervention
  Correlation between urine and serum levels of circulating parasite antigen and lesion resolution on MRI as a potential marker of treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Seth E O'Neal, MD MPH, Principal Investigator — Oregon Health and Science University; Hector H Garcia, MD PhD, Principal Investigator — Universidad Peruana Cayetano Heredia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient data for primary and secondary outcomes will be made available.
Time Frame: 6 months after trial completion
Access Criteria: Data access requests will be reviewed by the principal investigators. Requestors will be required to sign a Data Use Agreement.